CLINICAL TRIAL: NCT00879138
Title: A Double-blind, Placebo-controlled Dose Response Study to Investigate Pharmacodynamics and Pharmacokinetics of Single and Repeated Oral Doses of VA106483 in Elderly Male Subjects
Brief Title: Efficacy and Safety of VA106483 in Elderly Males
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vantia Ltd (Industry)
Collaborators: Veeda Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 483-001
Record Dates: First submitted 2009-02-18; First posted 2009-04-09 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Sugar pill
- VA106483 2 mg (Experimental)
  Interventions: Drug: VA106483
- VA106483 4 mg (Experimental)
  Interventions: Drug: VA106483
- VA106483 8 mg (Experimental)
  Interventions: Drug: VA106483

INTERVENTIONS:
Drug: VA106483
  Arms: VA106483 2 mg; VA106483 4 mg; VA106483 8 mg
Drug: Sugar pill
  Arms: Sugar pill

SUMMARY:
A double blind, placebo-controlled, dose ranging study in males over the age of 65, who have a history of nocturia. The study will investigate pharmacodynamic outcomes (urine volumes and osmolality, circulating coagulation factors and haemodynamics) and pharmacokinetics, of both single and multiple oral doses of VA106483 at three dose levels, under conditions of controlled hydration.

DETAILED DESCRIPTION:
VA106483 is a selective vasopressin V2 receptor agonist which is currently under development for the treatment of nocturia in males. This study examines the pharmacological action of VA106483 on markers of clinical efficacy (urine volumes and osmolality) and safety markers (coagulation factors and haemodynamics). The study will also assess the pharmacokinetics in the study population. The study design includes both cross-over and parallel phases so that pharmacodynamic and pharmacokinetic parameters can be assessed following both single and repeat dosing. Three dose levels will be given.

ELIGIBILITY:
Inclusion Criteria:

* Males 65 years and above with history of nocturia

Exclusion Criteria:

* Any clinically significant concomitant medical disease, condition or abnormal laboratory test result
* Participation in any other clinical study within 30 days
* Intake of non-prescription medication within 14 days

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic profile of VA106483

SECONDARY OUTCOMES:
Pharmacokinetic profile of VA106483
Safety and tolerability of VA106483

CONTACTS AND LOCATIONS:
Locations (1):
- Veeda Clinical Research, Plymouth, United Kingdom